CLINICAL TRIAL: NCT02161536
Title: Evaluation of the Performance of the Motus Cleansing System
Acronym: MSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Motus GI Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: CP-MCC-SA-0214
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Results first posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2017-03

CONDITIONS: Colonoscopy Procedure

STUDY DESIGN:
Intervention Model Description: Bowel cleansing level was evaluated by using the Boston Bowel Preparation Score (BBPS) at baseline and after the use of the Motus Cleansing System.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motus CleanC System (Experimental): Colonoscopy with Motus CleanC Syetem - Device Rev 2.0 ,enrolled under protocol Rev 3.0
  Interventions: Device: Motus Cleansing System
- Motus Cleansing System Rev 2.5 (Experimental): Colonoscopy with MCS Rev 2.5,enrolled under protocol Rev 4.0
  Interventions: Device: Motus Cleansing System
- Motus Cleansing System Rev 3.0 (Experimental): Colonoscopy with MCS Rev 3.0,enrolled under protocol Rev 5.0
  Interventions: Device: Motus Cleansing System

INTERVENTIONS:
Device: Motus Cleansing System
  Other Names: Motus CleanC

SUMMARY:
The purpose of this study is evaluate the Motus GI Colon Cleansing system performance.

DETAILED DESCRIPTION:
Subjects indicate for colonoscopy procedure undergo a limited bowel preparation including 20 mg Bisacodyl (4*4 tables of 5 mg each) in split dose undergo standard colonoscopy with MCS.

following the procedure 2 follow-up call were conducted at 48 hours and 14 days after to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in the age range of 18-75 years
* Subjects with BMI within the range of 18.5-35
* Subject is willing to sign informed consent form

Exclusion Criteria:

* Active or severe IBD
* Subjects with severe diverticulitis \ diverticular disease (known or detected)
* Known or detected colonic stenosis
* Known or detected bowel obstruction
* History of prior colon surgery
* ASA≥IV (sever systemic disease)
* Sever Renal insufficiency
* Sever Liver insufficiency
* Contraindication for "colonoscopy" anesthesia \ sedation \ prep agent pregnancy
* Subjects with altered mental status/inability to provide informed consent
* Subject has a condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound the study results, or may interfere significantly

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravit Peled, Study Director — Motus GI Technologies Ltd.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 3 phases:
  Phase 1 - enrolled 6 subjects using Rev 2.0 of the device Phase 2 - enrolled 21 subjects using Rev 2.5 of the device Phase 3 - enrolled 20 subjects using Rev 3.0 of the device
Pre-assignment Details: Patients had to follow a specific bowel preparation in order to mimic poor bowel preparation:
  Arm 1: start clear liquid diet 24 hours prior to the procedure Arm 2: start clear liquid diet 24 hours prior to the procedure Arm 3: start clear liquid diet 18 hours prior to the procedure along with 4 tables of 5 mg Bisacodyl in split dose
Groups:
- Motus CleanC Syetem Rev 2.0: 6 subjects used the second version of the device
- Motus Cleansing System Rev 2.5: 21 subjects enrolled under protocol Rev 4.0 , had a standard colonoscopy procedure with Motus Cleansing System Rev 2.5
- Motus Cleansing System Rev 3.0: 20 subjects enrolled under protocol Rev 5.0 , had a standard colonoscopy procedure with Motus Cleansing System Rev 3.0
Period: Overall Study
Arm/Group | Motus CleanC Syetem Rev 2.0 | Motus Cleansing System Rev 2.5 | Motus Cleansing System Rev 3.0
Started | 6 | 21 | 20
Completed | 6 | 21 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Motus CleanC System Rev 2.0: Motus CleanC System Rev 2.0
- Motus Cleansing System Rev 2.5: Motus Cleansing System Rev 2.5
- Motus Cleansing System Rev 3.0: Motus Cleansing System Rev 3.0
- Total: Total of all reporting groups
Arm/Group | Motus CleanC System Rev 2.0 | Motus Cleansing System Rev 2.5 | Motus Cleansing System Rev 3.0 | Total
Number analyzed (Participants) | 6 | 21 | 20 | 47
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 48 (8.7) | 49.2 (11.6) | 54.7 (6.6) | 51.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 8 | 18
  Male | 3 | 14 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: The Count and Percentage of Subjects Had Adequate Bowel Preparation After the Use of Motus Cleansing Stystem
Description: The number of subjects had adequate bowel preparation after the use of Motus Cleansing System (i.e., all colon segments have BBPS>=2) .
  Each colon segment was graded by using the Boston Bowel Preparation Score index before ( at baseline) and after the cleansing of the bowel by using the Motus Cleansing System.
Time Frame: Following the colonoscopic procedure- Up to 24 hours.
Population: subjects had adequate bowel preparation after the use of Motus Cleansing System (i.e., all colon segments have BBPS>=2)
Measure: Count of Participants; unit: Participants
Groups:
- Motus CleanC System: Colonoscopy with Motus CleanC Syetem - Device Rev 2.0 ,enrolled under protocol Rev 3.0
  Motus Cleansing System
- Motus Cleansing System Rev 2.5: Colonoscopy with MCS Rev 2.5,enrolled under protocol Rev 4.0
  Motus Cleansing System
- Motus Cleansing System Rev 3.0: Colonoscopy with MCS Rev 3.0,enrolled under protocol Rev 5.0
  Motus Cleansing System
Arm/Group | Motus CleanC System | Motus Cleansing System Rev 2.5 | Motus Cleansing System Rev 3.0
Number analyzed (Participants) | 6 | 21 | 20
Participants | 6 | 20 | 20

ADVERSE EVENTS:
Arm/Group | Motus CleanC Syetem Rev 2.0 | Motus Cleansing System Rev 2.5 | Motus Cleansing System Rev 3.0
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 3/6 | 2/21 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motus CleanC Syetem Rev 2.0 (N=6) | Motus Cleansing System Rev 2.5 (N=21) | Motus Cleansing System Rev 3.0 (N=20)
Bowel perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — The head design comprises flexible balcony-like in the tip which was beyond the scope's field of view, are suspected as the cause for the perforation. The event was resolved with a scar as a residual effect.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motus CleanC Syetem Rev 2.0 (N=6) | Motus Cleansing System Rev 2.5 (N=21) | Motus Cleansing System Rev 3.0 (N=20)
Laceration (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) — mild laceration resolved with no clinical sequelae within two days
Erosion (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) — mild erosion resolved with no clinical sequelae
Submucosal Hematoma (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) — mild Hematoma resolved with no clinical sequelae

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No